CLINICAL TRIAL: NCT07256080
Title: A Sham-Controlled Cross-Over Study Examining the Effects of Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) on Cognitive Performance and Gender Differences in Healthy Adults
Brief Title: Effects of Transcutaneous Auricular Vagus Nerve Stimulation on Cognitive Performance and Sex Differences
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Yara Atef Skout, Principal investigator, Bahçeşehir University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 61351342/020-93
Record Dates: First submitted 2025-11-18; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Assessment; Cognition; taVNS; Vagus Nerve Stimulation; Executive Functions; Healthy Participants; Neuromodulation; Sex Differences

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to whether they receive active or sham stimulation. Outcome measures (CogniFit, HRV, STAI, PSS) are automated or self-administered; outcome assessors will therefore be blinded to condition. The investigator applying stimulation will not be blinded due to device setup requirements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active taVNS Stimulation (Experimental): Active taVNS will be applied bilaterally to the cymba conchae and tragus regions using the VaguStim device. Stimulation will follow standard parameters used in cognitive studies to minimize cardiac side effects. Parameters: biphasic waveform, 25 Hz frequency, 250 μs pulse width, and intensity individually adjusted below the sensory threshold (0.5-4 mA). Each session will last 20 minutes.
  Interventions: Device: Active taVNS
- Sham Stimulation (Sham Comparator): For the sham condition, electrodes will be placed on the earlobe bilaterally, an area not innervated by the vagus nerve, using the same device and parameter settings but without delivering active stimulation. This setup controls for placebo effects.
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Active taVNS — Active taVNS will be delivered bilaterally to the cymba conchae and tragus regions using the VaguStim device. Stimulation parameters follow cognitive-neuroscience standards to minimize cardiac side effects: biphasic waveform, 25 Hz frequency, 250 μs pulse width, and intensity individually adjusted below the sensory threshold (0.5-4 mA). Each stimulation session lasts 20 minutes.
  This intervention corresponds to the Active taVNS Stimulation arm.
  Arms: Active taVNS Stimulation
Device: Sham Stimulation — Sham stimulation will be delivered using the same VaguStim device, but electrodes will be placed bilaterally on the earlobe, an area not innervated by the vagus nerve. Device parameters will be set to match the active condition, but no true vagus nerve stimulation is delivered. This procedure controls for placebo and participant expectancy effects.
  This intervention corresponds to the Sham Stimulation arm.
  Arms: Sham Stimulation

SUMMARY:
This study investigates the effects of transcutaneous auricular vagus nerve stimulation (taVNS) on cognitive performance in healthy adults. The study uses a sham-controlled, cross-over design in which each participant receives both active taVNS and sham stimulation in separate sessions. Each participant completes both conditions (active and sham) in a randomized order using a crossover design. Cognitive performance will be assessed before and after each session using standardized tests. The study also explores whether males and females respond differently to taVNS, in order to identify potential sex-related differences in cognitive outcomes.

DETAILED DESCRIPTION:
This randomized, sham-controlled cross-over study investigates the effects of transcutaneous auricular vagus nerve stimulation (taVNS) on cognitive performance, autonomic activity, and psychological state in healthy young adults, with specific attention to sex differences. Because hormonal fluctuations may influence vagal tone and cognitive outcomes, female participants are required to complete their stimulation sessions during the follicular phase (Day 5-10) of the menstrual cycle. Male participants follow the same protocol without timing restrictions.

The study consists of three laboratory visits, scheduled one week apart.

Visit 1 (Baseline Assessments):

Participants provide informed consent and complete a demographic questionnaire, menstrual-cycle verification (for female participants), the Montreal Cognitive Assessment (MoCA), and baseline psychological questionnaires including the State-Trait Anxiety Inventory (STAI) and the Perceived Stress Scale (PSS). Baseline cognitive performance is measured using the CogniFit digital battery.

Visits 2 and 3 (Randomized Cross-Over Stimulation Sessions):

Participants undergo active taVNS and sham stimulation in randomized order. At the beginning of each visit, heart rate variability (HRV) is recorded for 5 minutes before stimulation to establish a resting baseline. Stimulation is applied for 20 minutes using the VaguStim device. Immediately after stimulation, HRV is recorded again for 5 additional minutes, followed by completion of a side-effect questionnaire documenting any sensations or adverse reactions. Following that, participants complete the STAI and PSS questionnaires to assess post-stimulation psychological state.Cognitive performance is then reassessed using the CogniFit digital battery.

This cross-over design enables within-subject comparison between active and sham stimulation and provides the structure needed to examine potential sex-related differences in autonomic, cognitive, and psychological responses to taVNS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults aged 18-30 years
* Ability to provide informed consent
* Right-handed participants (to reduce variability in cognitive performance)
* Normal or corrected-to-normal vision and hearing
* Female participants tested during the follicular phase of the menstrual cycle (days 5-10) to minimize hormonal effects on cognition and vagal tone

Exclusion Criteria:

* History of neurological or psychiatric disorders
* Cardiovascular disease
* Use of psychoactive medications
* Substance dependence, including alcohol, illicit drugs, or nicotine
* Pregnancy or breastfeeding
* Skin conditions or ear anomalies that interfere with electrode placement
* Metal implants in the head or neck region
* History of epilepsy or migraine

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
CogniFit Digital Battery | Day 1 (Visit 1 baseline), Day 8 (Visit 2), and Day 15 (Visit 3) Cognitive testing will occur after stimulation on Day 8 and Day 15.
  Cognitive performance will be evaluated using the CogniFit digital cognitive battery, which assesses multiple cognitive domains including attention, working memory, executive functions, and processing speed.
  The battery will be administered once at baseline (Visit 1). It will be administered again immediately after Active stimulation in Visit 2 and immediately after Sham stimulation in Visit 3.
  Changes in cognitive scores between baseline and post-stimulation sessions will be compared to determine the acute cognitive effects of active vs. sham taVNS.

SECONDARY OUTCOMES:
Heart Rate Variability (HRV) | Day 8 (Visit 2): 5 minutes before stimulation and 5 minutes after stimulation. Day 15 (Visit 3): 5 minutes before stimulation and 5 minutes after stimulation.
  Heart rate variability will be assessed using the Polar H10 chest strap or another validated portable HRV device widely used in research. Five-minute recordings will be obtained during resting state and during stimulation. Time-domain parameters (RMSSD, SDNN) and frequency-domain parameters (LF/HF ratio) will be analyzed.
Perceived Stress Levels (PSS) | Day 1 (Visit 1 baseline), Day 8 (Visit 2 after stimulation), and Day 15 (Visit 3 after stimulation).
  The Perceived Stress Scale (PSS) will assess participants' perceived stress levels over the past month. Higher scores indicate higher perceived stress.
State and Trait Anxiety (STAI) | Day 1 (Visit 1 baseline), Day 8 (Visit 2 after stimulation), and Day 15 (Visit 3 after stimulation).
  The State-Trait Anxiety Inventory (STAI) will measure acute state anxiety (STAI-S) and general trait anxiety (STAI-T).
Self-Reported Side Effects | Day 8 (Visit 2 after stimulation) and Day 15 (Visit 3 after stimulation)
  A researcher-developed side-effects questionnaire will be used to record any discomfort, tingling, dizziness, or other adverse effects following stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Veysel Ozden, Study Chair — Bahçeşehir University

IPD SHARING:
Plan to Share IPD: No